CLINICAL TRIAL: NCT03900741
Title: Guided Bone Regeneration of Peri-implant Defects Comparing Submerged Versus Non-submerged Healing: a Randomized Controlled Clinical Trial
Brief Title: Guided Bone Regeneration of Peri-implant Defects Comparing Submerged Versus Non-submerged Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ana Molina Villar (Other)
Responsible Party: Sponsor-Investigator, Ana Molina Villar, Investigator, Universidad Complutense de Madrid
Organization: Universidad Complutense de Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18/575-R_X
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Peri-Implantitis
Keywords: Peri-Implantitis; Peri-Implant Diseases; Bone Regeneration; Submerged Healing; Non-Submerged Healing; Dental Implants
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Submerged healing (Experimental): Bone regeneration of peri-implantitis defects following a submerged healing
  Interventions: Procedure: Submerged healing
- Non-submerged healing (Active Comparator): Bone regeneration of peri-implantitis defects following a non-submerged healing
  Interventions: Procedure: Non-submerged healing

INTERVENTIONS:
Procedure: Submerged healing — Bone regeneration of peri-implantitis defects using a bone xenograft and a resorbable collagen membrane, with flap suturing using a submerged healing protocol
  Arms: Submerged healing
Procedure: Non-submerged healing — Bone regeneration of peri-implantitis defects using a bone xenograft and a resorbable collagen membrane, with flap suturing using a non-submerged healing protocol
  Arms: Non-submerged healing

SUMMARY:
Objective: the objective of the present randomized clinical trial is to compare changes in radiographic peri-implant bone defect fill after regeneration of peri-implant intrabony defects with a submerged versus a non-submerged protocol.

Material and Methods: this project is a randomized controlled clinical trial, double blind, with a parallel groups design. Thirty-six patients presenting with peri-implantitis subsidiary of regenerative treatment will be recruited. After subjects have been given informed consent, they will be randomized to test or control group. All patients will undergo a session of non-surgical peri-implantitis therapy consisting on prostheses removal and implant debridement with ultrasounds, curettes and air-abrasive under local anaesthesia. Patients in test group will have their prostheses removed and the mucosa surrounding the affected implants will be let heal covering the implants, while patients in control group will have their prostheses installed again after the non-surgical therapy. Six to eight weeks later, all subjects will undergo regenerative treatment with the use of a bone substitute, a collagen membrane and fixation pins, and in control group tissues will heal following the non-submerged protocol, meanwhile subjects in test group will undergo submerged healing. Six months later, subjects in test group will have their prostheses reconnected to the regenerated implants. All patients will undergo periodontal and peri-implant maintenance therapy every three months during follow-up. Radiographic assessment of vertical bone level changes (primary outcome), clinical status of peri-implant tissues, changes in soft tissues margin, patient related outcomes and adverse events will be assessed at 3, 6 and 12 months after peri-implantitis regenerative surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of peri-implantitis requiring surgical therapy
* The periapical radiographic study demonstrates an intra-bony component greater than 3 mm at the affected implant
* There is at least 2 mm of keratinized mucosa around the affected implant
* Intrasurgically, peri-implant defects must be type Ia, Ib, Ic and Ie (according to Schwarz et al. 2007)
* Affected implants must be two-piece implants to allow for the submerged protocol
* Affected implant supported restorations must be screw-retained or cemented, and should allow for prostheses removal

Exclusion Criteria:

* Patients with untreated periodontitis
* Medical conditions requiring prolonged use of steroids and/or medications that can interfere with bone metabolism
* Metabolic disorders such as osteoporosis
* History of uncontrolled endocrine disorders
* History of leukocyte dysfunction and deficiencies
* History of immunodeficiency syndromes
* History of neoplastic disease requiring the use of radiation of chemotherapy
* History of renal failure
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Alcoholism or drug abuse
* Smokers of more than 10 cigarettes per day, cigar equivalents or tobacco chewers
* Any other condition or circumstance that, in the opinion of the investigator, would prevent completion of study participation or interfere with the analysis of the study results, such as history of non-compliance or unreliability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Changes in radiographic bone fill | Baseline, 3 months, 6 months and 12 months post-surgery
  Changes in radiographic bone fill measured from the implant shoulder to the first bone to implant contact with ImageJ software, in parallelized periapical x-rays with individual silicone bite blocks

SECONDARY OUTCOMES:
Changes in pocket probing depth | At baseline, after non-surgical therapy, 6 months and 12 months post-surgery
  Depth of the peri-implant sulcus/pocket measured in millimeters with a 15-UNC (University of North Carolina) periodontal probe, at six sites per implant without the crown
Changes in bone probing depth | At baseline, after non-surgical therapy and 12 months post-surgery
  Distance from the mucosal margin to the peri-implant bone measured in millimeters with a 15-UNC (University of North Carolina) periodontal probe under local anesthesia, at six sites per implant without the crown
Changes in modified plaque index | At baseline, after non-surgical therapy, 6 months and 12 months post-surgery
  Presence or absence of plaque assessed at six sites per tooth/implant in the whole mouth, excluding third molars
Changes in full mouth bleeding scores | At baseline, after non-surgical therapy, 6 months and 12 months post-surgery
  Presence or absence of bleeding after probing with a 15-UNC (University of North Carolina) periodontal probe, assessed at six sites per tooth/implant in the whole mouth, excluding third molars. The presence of bleeding in each site will be scored 1, and the absence of bleeding will be scored 0. Full mouth bleeding score will be expressed in percentage and calculated as follows: number of sites bleeding / number of sites explored ^ 100
Soft tissue healing scores | 1 week, 2 weeks and 4 weeks post-surgery
  Extent of soft tissue healing after surgery following Landry et al. Healing Index (1988):
  * Healing index 1 - Very Poor
  * Healing index 2 - Poor
  * Healing index 3 - Good
  * Healing index 4 - Very good
  * Healing index 5 - Excellent
Pain assessment | 1 week, 2 weeks and 4 weeks post-surgery
  Participants´ subjective pain assessed using a Visual Analogue Scale (VAS) with ratings from 0-10, whereof 0 = no pain and 10 = very intense.
Oral Health Impact Profile (OHIP-14) | Baseline, 3 months, 6 months and 12 months post-surgery
  Self-reported dysfunction, discomfort and disability attributed to the participants´ oral condition
Adverse events´ occurrence | Up to 12 months post-surgery
  Occurrence of any untoward, undesired or unplanned event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a subject participant in the clinical investigation. The event does not nee to be casually related to the cliinical investigation

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, MD DDS DrMed, Principal Investigator — University Complutense of Madrid
Locations (1):
- Dental School, University Complutense of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No